## **COVER PAGE**

## The Dedicated African American Dad Study NCT number-NCT02412748

Document date- July 6, 2018

**Mother Telephone Informed Consent Document** 

ORA: 14022704-IRB01-CR03 Date IRB Approved: 7/6/2017 Expiration Date: 7/6/2018

## The African American Non-resident Fatherhood Program Mother/Guardian Telephone Script

Hi, my name is [state your name]. I'm working on a research study called the D.A.A.D. Study to help African American fathers be the best fathers they can be when they live in a different home than their children. Is this a good time for you to talk?

- If yes, continue with script below.
- ❖ If no, ask to set up another time to talk with them about the study.

We are inviting you to take part in this study because the father of a child in your care signed up to participate. He thought you would be open to supporting his participation. This study is being conducted by Dr. Wrenetha Julion from Rush University College of Nursing. Have you already received the information letter and consent forms for the study?

| *** | If yes, continue below with the purpose of the study and what they will need to do to |
|---|---|
| | participate. |
| <b>*</b> | If no, but the potential subject is interested in hearing more about the study now, |
| | ☐ Tell them about the purpose of the study |
| | ☐ Tell them what they will need to do to participate. |
| | □ Arrange to send the information letter and consent forms by mail, email or fax. |
| | ☐ Schedule a time to talk to them again for consenting and interview either over the phone |
| | or in person. |
| | ☐ Verify address and/or email address to send consent forms: |
| | 2 |
| | Ammuorrad # |
| | 3 ADDroved # 3 |

If not, interested in being part of the study, thank them for their time.

The purpose of this study is to test two different programs. One program is about fatherhood and the other program is about financial planning.

If you decide to take part in this study, you will be asked to answer some questions about the child, the time they spend with their father and your co-parenting relationship with the child's father. We plan to have 180 fathers and 180 mothers or guardians take part in this study. Your participation is completely voluntary. We will ask you to complete the interview before the program starts, at the end of the 12-week program, and again 3 months after the program ends. Your entire time in the study will last about 9 months. You will be paid \$40 each time you complete the interview. For the first interview, it will take about an hour to complete the consent process and do the interview. For the second and third interviews, it will take about 30-45 minutes. Do you have any questions about the study? Are you interested in participating now over the phone or in person?

- ❖ If now over the phone, answer any questions they may have. Then, complete the interview.
- If the mother/guardian does not have time right now, schedule an appointment either on the phone or in person to obtain the consent and conduct the interview.

 Version Date: 12/09/2014

| ☐ Verify the <b>best telephone number</b> to cond | luct the telephone interview: |
|---|---|
| Phone #: | |
| ☐ Set up the telephone interview: | |
| Date & Time: | |
| <u>OR</u> | |
| Set up the in-person interview: | |
| Date & Time: | |
| Address: | |
| this call go over the consent and HIPAA form. After verify that the mother/guardian understands the form the risks and benefits of the study? The risks and benefits of the study? The alternatives to participating? Their rights while participating in the study? Who is sponsoring the study? Who they should contact with any quest will do to protect their confider. Their rights regarding protected health Verify the following: Do you have any questions? [Answer any questions.] Do you agree to participate in this study? Yes: Document Research and HIPAA consent below and | er going over the consent and HIPAA forms, ollowing: ddy tions or concerns about the study? ntiality? information |
| Informed Consent for Research HIPAA Consent | 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 |
| No: Thank them for their time. | Appear |
| Name of Subject: | |
| [Verify correct spelling of name] | |
| Person Obtaining Consent I have read this form to the subject. An explanation of the subject were solicited and answered to the subject's satisdemonstrated comprehension of the information. The successent to participate in this study. | sfaction. In my judgment, the subject has |
| Name and Title (Print) | |
| | Version Date: 12/09/2014 |

ORA: 14022704-IRB01-CR03 Date IRB Approved: 7/6/2017 Expiration Date: 7/6/2018

 Version Date: 1

ORA: 14022704-IRB01-CR03 Date IRB Approved: 7/6/2017 Expiration Date: 7/6/2018 Signature of Person Obtaining Consent Date

 Version Date: 12/09/2014